CLINICAL TRIAL: NCT03360422
Title: Advancing New Computer-based Health Outcomes Regarding Sexual Behavior(ANCHORS) Study: UH2 Project
Brief Title: ANCHORS Study: UH2 Project
Acronym: ANCHORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB201701367 N; UH2AA026214-01 (NIH)
Record Dates: First submitted 2017-11-20; First posted 2017-12-04 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: HIV-1-infection
Keywords: MSM, young adult
MeSH Terms: interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Survey group (Active Comparator): Collect alcohol and sexual activity data via web survey from 683 young MSM to yield normative data for the alcohol and HIV preventive intervention in a follow-up study
  Interventions: Other: Survey
- Focus Group (Active Comparator): 30 young MSM who drink regularly to inform the content of the alcohol and HIV preventive intervention tested in the UH3 phase and ensure the intervention is culturally appropriate for MSM.
  Interventions: Other: Survey; Other: Focus Group
- Usability Study (Active Comparator): 10 young adult MSM will test the mobile intervention in development for 30 days in order to establish usability, acceptability and correct any functionality issues.
  Interventions: Other: Survey; Other: Usability study

INTERVENTIONS:
Other: Survey — Respondents meeting inclusion criteria will be informed they were selected for the longer survey and continue to the survey. Upon completion, the survey will generate a study identification (ID) that respondents will provide to study staff with additional contact information via phone, text or email to be compensated
Other: Focus Group — After informed consent, participants will complete the web-based intervention component in development. Afterward, participants will be engaged by an experienced facilitator in a discussion of aspects of the intervention they liked and disliked and suggestions they have for enhancing its cultural appropriateness to young MSM.
  Arms: Focus Group
Other: Usability study — After informed consent, participants will utilize the mobile intervention in development for 30 days to establish usability, acceptability and correct any functionality issues.
  Arms: Usability Study

SUMMARY:
According to the National HIV/AIDS Strategy, men who have sex with men (MSM), young adults, Black and Latino men and people in the Southern U.S. are at highest HIV risk and should be targeted with cost-effective, scalable interventions. The study team propose a synergistic mobile intervention to reduce alcohol and HIV risk in young adult MSM that combines 3 efficacious approaches.

DETAILED DESCRIPTION:
New prevention efforts must address alcohol and HIV and be directed to the highest-risk groups. While interventions have targeted MSM, few have targeted young MSM specifically. Young people and MSM bring particular challenges. Thus, it is important that prevention be targeted to them and developed with their input. To that end, the goal of this project is to lay the groundwork for a synergistic, mobile intervention to reduce alcohol use and risky sex and prevent HIV among young adult MSM. This research study is made up of three related sub-projects: 1) a web-based survey; 2) a series of focus groups and 3) a small, preliminary acceptability and usability to study to test the mobile intervention. The proposed intervention to be tested on a preliminary basis in this study combines brief motivational intervention with daily interactive voice response (IVR) monitoring including personalized feedback. Ultimately, this combined intervention will also include pre-exposure prophylaxis (PrEP), however there will be no medication in this particular study. Each of these components has efficacy in enhancing treatment adherence, reducing alcohol and/or HIV risk but requires other interventions to maximize its potential benefit. Combining them will capitalize on the strength of each, leading to a higher impact alcohol and HIV preventive intervention.

ELIGIBILITY:
Inclusion Criteria:

Web-survey:

* Male sex
* Ages 18-30
* Ability to read and write English
* 1 or more instances of sexual activity with another man in the past 3 months
* HIV Negative

Focus group:

* 18-35
* All other inclusion criteria will be the same as the web survey

Usability phase:

* 5 or more drinks in a day in the past month
* Past-month intercourse with another man without a condom
* Willingness to try PrEP, but have never tried it before

Exclusion Criteria:

Web Screen:

- No subject may have lifetime use of PrEP

Focus group:

* A current undergraduate or graduate student at any level in one of the 3 departments that make up the College of Health and Human Performance (HHP) at the University of Florida (UF), where Dr. Leeman's faculty appointment is.
* Do not want to engage in open discussion regarding substance use or sexual activity/orientation in a group setting. It will be possible for participants to contribute to focus group discussions without providing detailed information about their own substance use or sexual activity, however focus group participants must have a degree of openness to discussing these topics with others. These groups will take place with 6-7 other people and some people may be made uncomfortable by the discussions that may take place with regard to participants' drinking, substance use or sexual behavior.
* Not willing to be recorded via an electronic recording device

Usability phase:

* No subject may have lifetime use of PrEP
* Those who do not wish to provide a reliable phone number will be excluded

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 673 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Leeman, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who enrolled in a focus group/individual interview and the usability study were a subset of those who completed the survey
Pre-assignment Details: Provision of insufficient data to be considered a valid participant
Groups:
- Young Adult Men Who Have Sex With Men: 18-30 young men who have sex with men
Period: Survey
Arm/Group | Young Adult Men Who Have Sex With Men
Started | 673
Completed | 673
Not Completed | 0
Period: Focus Group/Individual Interview
Arm/Group | Young Adult Men Who Have Sex With Men
Started | 24
Completed | 24
Not Completed | 0
Period: Usability Study
Arm/Group | Young Adult Men Who Have Sex With Men
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Young Adult Men Who Have Sex With Men: 18-30 year old men who have sex with men residing in the Southern United States
Arm/Group | Young Adult Men Who Have Sex With Men
Number analyzed (Participants) | 673
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 673
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.77 (3.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 673
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 153
  Not Hispanic or Latino | 509
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 117
  White | 458
  More than one race | 41
  Unknown or Not Reported | 24
Region of Enrollment [Number; unit: participants]
  United States | 673

OUTCOME MEASURES:

1. Primary Outcome: Quantity of Alcohol Consumption
Description: Determine levels of alcohol consumption in study population
Time Frame: Retrospective self-report over the past month
Measure: Mean (Standard Deviation); unit: drinks
Groups:
- Survey Group: Collect alcohol and sexual activity data via web survey from 673 young MSM to yield normative data for the alcohol and HIV preventive intervention in a follow-up study
  Survey: Respondents meeting inclusion criteria will be informed they were selected for the longer survey and continue to the survey. Upon completion, the survey will generate a study identification (ID) that respondents will provide to study staff with additional contact information via phone, text or email to be compensated
- Focus Group/Individual Interview: 24 young MSM who drink regularly to inform the content of the alcohol and HIV preventive intervention tested in the UH3 phase and ensure the intervention is culturally appropriate for MSM.
  Survey: Respondents meeting inclusion criteria will be informed they were selected for the longer survey and continue to the survey. Upon completion, the survey will generate a study identification (ID) that respondents will provide to study staff with additional contact information via phone, text or email to be compensated
  Focus Group: After informed consent, participants will complete the web-based intervention component in development. Afterward, participants will be engaged by an experienced facilitator in a discussion of aspects of the intervention they liked and disliked and suggestions they have for enhancing its cultural appropriateness to young MSM.
Arm/Group | Survey Group | Focus Group/Individual Interview | Usability Study
Number analyzed (Participants) | 673 | 24 | 10
drinks | 11.38 (20.05) | 7.81 (7.80) | 4.78 (2.78)

2. Primary Outcome: High-risk Sexual Behavior: Condomless Sex
Description: Past month frequency of condomless sex
Time Frame: Retrospective self-report from past month on web survey
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Survey Group | Focus Group/Individual Interview | Usability Study
Number analyzed (Participants) | 673 | 24 | 10
events | 4.12 (6.92) | 2.22 (3.23) | 7.17 (9.39)

3. Primary Outcome: Study Participant Opinions on Acceptability of Intervention Content
Description: Participants in the usability study will report on the acceptability of the interactive voice response (IVR) system and the personalized feedback produced based on their IVR responses.
  On a modified System Usability Scale, participants in the usability study will report on the acceptability (i.e., perceived value, liking) of the interactive voice response (IVR) system and the personalized feedback produced based on their IVR responses. Items were rated on a 1-7 scale with higher scores indicating greater usability. The acceptability subscale is made up of 5 items. The score reported below is the mean of these five items.
Time Frame: Up to one month
Population: Acceptability was assessed only among participants in the usability study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survey Group | Focus Group/Individual Interview | Usability Study
Number analyzed (Participants) | 0 | 0 | 10
score on a scale |  |  | 5.50 (1.51)

4. Primary Outcome: Study Participant Opinions on Usability of Intervention Content
Description: On a modified System Usability Scale, participants in the usability study will report on the usability of the interactive voice response (IVR) system and the personalized feedback produced based on their IVR responses. Items were rated on a 1-7 scale with higher scores indicating greater usability. The usability subscale is made up of 4 items. The score reported below is the mean of these four items.
Time Frame: Up to 1 month
Population: Acceptability and usability data were collected only from the usability study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survey Group | Focus Group/Individual Interview | Usability Study
Number analyzed (Participants) | 0 | 0 | 10
score on a scale |  |  | 6.40 (0.70)

5. Primary Outcome: High-risk Sexual Behavior: Sexual Activity During/After Alcohol Use
Description: Past month frequency of alcohol use before or during oral, anal and/or vaginal sex
Time Frame: Past month on a self-report survey
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Survey Group | Focus Group/Individual Interview | Usability Study
Number analyzed (Participants) | 673 | 24 | 10
events | 2.88 (5.16) | 2.13 (3.49) | 1.50 (1.05)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse event data were collected from usability study participants using the SAFTEE. Adverse events were not monitored in the survey or focus group/interviews. Surveys were completed via the web. Focus groups/interviews occurred within a single session of about an hour to an hour and a half in which participants answered questions, thus adverse events were not possible in these parts of the study.
Arm/Group | Survey Group | Focus Group/Individual Interview | Usability Study
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT03360422/Prot_SAP_001.pdf
  • Informed Consent Form (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT03360422/ICF_000.pdf